CLINICAL TRIAL: NCT04058847
Title: Danish Evaluation of Your Heart Forecast. A Study Among Danish General Practitioners and Patients in the Blood Pressure Control Program.
Brief Title: Danish Evaluation of Your Heart Forecast.
Acronym: DANY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other); Odense Patient Data Explorative Network (Other); ENIGMA Solutions Limited (Unknown); Lilly & Herbert Hansens Foundation (Unknown); The A. P. Møller and Chastine McKinney Møller Foundation (Unknown)
Responsible Party: Principal Investigator, Anders Elkær Jensen, Medical doctor, Principal Investigator, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-20170206
Record Dates: First submitted 2018-10-26; First posted 2019-08-16 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Risk Communication; Cardiovascular Risk Factor
Keywords: Risk communication; CVD-risk; General practice; Primary care; Visual communication; Interactive communication; Cardiovascular risk

STUDY DESIGN:
Intervention Model Description: Cluster-randomised clinical trial with 1 year follow up. The general practitioners are randomised into an intervention group and a control group. Participants automatically follow their general practitioner into the allocated group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Use of Your Heart Forecast and an e-mail follow up-program.
  Interventions: Other: Your Heart Forecast
- Control (No Intervention): The control group uses standard regime (business as usual).

INTERVENTIONS:
Other: Your Heart Forecast — 1 year follow up with Your Heart Forecast and a follow-up email every 2 weeks.
  Arms: Intervention

SUMMARY:
Under 50% of patients diagnosed with hypertension and treated in general practice, have reached a blood pressure within the recommended levels of the national guideline. Compliance is the main problem for these patients, but effective tools for increasing patient compliance are missing. The objective is to evaluate the risk-assessment and risk-communication tool: "Your Heart Forecast", to see if it can improve patient compliance, health literacy and empowerment.

Patients will be followed in a cluster-randomised controlled trial in the setting of general practice, using surveys at inclusion and after 6 and 12 months. Besides surveys, the participants' blood pressure will be measured as a hard outcome and data will be drawn from various patient databases. After 6 months, qualitative interviews will be conducted, with a subgroup of patients from the intervention group.

It is expected to find whether the use of Your Heart Forecast can lower patients' blood pressure and/or increase their compliance, health literacy and empowerment. The aim is to show if an increase in general health literacy and patient empowerment, as measured by Patient Activation Measure(PAM13) can be seen.

The investigators hope to reveal whether this software can improve patient compliance and thereby be a reasonable tool to implement in the national blood pressure control program. In further studies, it should be shown if the cost of using this program is far less than expenses for hospitalisation due to complications and comorbidity to hypertension.

DETAILED DESCRIPTION:
The project description has been shortened to fit the format of clinicaltrials.gov.

Background:

To improve communication of risk messages, they must be communicated in a way that is understandable and relevant to the patient. Every individual is different and therefore communication tools must be personalised and easy to understand. This is important as low health literacy is present among close to half of the European population and is associated with poor health outcomes, low self-management and underestimation of personal Cardiovascular Disease (CVD) risk. Since the risk of CVD is the product of a complex combination of multiple individual risk factors, there is a need for communicating complex information in an easily understandable way. Several tools for calculating and communicating CVD risk have been developed, but rigorous testing of their communicative effects is lacking.

Inadequately controlled blood pressure is associated with an increased risk of CVD, and more frequent contacts with GPs. Intention to change behaviour is related to the patients' perception of risk. Consequently, better ways for GPs to communicate CVD risks and motivate patients for risk-reducing strategies are warranted. Efficient communication requires information to be presented in formats that encourage decision-makers, i.e. patients, to automatically extract specific meanings or overall messages. Use of graphical illustrations with distinct features has previously been shown to be an effective and user-friendly tool to communicate risk, especially to people with limited health literacy. A visual decision aid could be a way to improve the blood pressure consultations and to assure that GPs are supported to provide patients with the relevant information. It is suggested that using a decision aid will also systematise the consultation and make it more reproducible.

The present study will use the internet-based risk communication tool Your Heart Forecast (YHF) to evaluate, whether it can influence patients' understanding of risk and treatment adherence. This will be done paying special attention to patients' blood pressure, lipid levels, empowerment and health literacy. The rationale behind the tool is to help improve patient-doctor interaction and communication so that the patient can gain an improved understanding of his/her CVD risk, and the modifiability of risk. Patients with hypertension have been chosen as a case study since high blood pressure is one of the main modifiable risk factors for CVD, as opposed to i.e. age, gender, ethnicity and family history.

YHF is a risk-communication tool, which communicates CVD risks as personalised, interactive and dynamic visual graphs. Following input from personal health-related data, the GP can, by using YHF, interactively guide the patient through:

* Their currently predicted 5-year absolute CVD risk
* The age at which they would achieve their currently predicted CVD risk if they had ideal/achievable risk factor control (the heart age)
* Their predicted CVD risk as they get older (the heart forecast)
* Their future CVD risk if their current risk factors are improved. As it has previously been demonstrated that single event interventions do not have an effect if not followed up, YHF will be introduced in a package deal. YHF will function as the primary intervention and repeated reminders via e-mail will be the secondary component. Patients in the intervention group will, after the consultation with the GP, receive emails every other week, as part of a general health literacy educational program.

Aim:

The aim is to evaluate the effect of using the YHF visual communication tool on changes in blood pressure and adherence to CVD preventive medications. Further, by means of questionnaires, it is the aim to study whether changes in health-literacy, adherence, patient empowerment and risk communication are associated with changes in blood pressure, lipid levels and/or lifestyle choices. By means of qualitative interviews, it will be investigated whether the use of the program heightens motivation, increases awareness of risk or creates unwarranted effects like causing the patients to be anxious.

Primary research question:

• Will the introduction of YHF during an annual blood pressure control consultation lead to improved general health literacy, improved medication adherence and empowerment after 12 months?

Secondary research questions:

1. Will blood pressure be reduced among patients in the intervention group compared to the control group after 12 months?
2. Will lower health literacy and/or low empowerment at baseline be associated with higher blood pressure at baseline?
3. Will health literacy and/or empowerment be improved after 6 and/or 12 months among patients enrolled in the intervention group?
4. Will increased health literacy and/or empowerment be associated with healthier lifestyle including diet, exercise and smoking habits after 12 months?
5. Will there be subjective feelings of increased motivation or sickening after introducing the intervention?
6. Will CVD risk be lower among patients in the intervention group compared to the control group after 12 months?

Methods

Trial design:

This study will use a mixed methods approach with a combination of a randomised controlled trial (RCT) and qualitative semi-structured interviews. The protocol has been developed using the SPIRIT checklist as a guideline.

Two pilot practices will be enrolled as if they were intervention practices. In these 2 practices, patients will be assessed 3-6 months before the project practices. A subgroup Q, of 5-15 patients from the pilot group, will be selected for qualitative interviews.

GPs in the control group, will not be introduced to YHF and will follow their patients in the blood pressure control program as usual.

Study population Participants All general practices in the Region of Southern Denmark will be invited to join the study. 30 GPs of those willing to participate, will, with due respect for geographical location and practice type, be representatively selected for participation.

Both incident and prevalent hypertensive patients will be included within an inclusion period of 6-12 months.

Sample size Sample size calculation is based on blood pressure as the primary outcome. For a two-sample pooled t-test of a normal mean difference with a two-sided significance level of 0.05, a sample size of 120 participants per group is required. This is to obtain a power of at least 90%, to detect a difference of 5 mmHg between the means at baseline and after 1 year. To adjust for expected drop-outs, 30 participants will be added per group and at least 300 patients will be enrolled in the trial. To account for cluster-effects when randomising on practice-level, the sample size will be further increased by 10-15% to reach 340 patients. More participants will be needed for subgroup analyses on sociodemographic and therefore, the aim is to reach a total of 600 participating patients. The pilot practices will provide information regarding the prevalence of patients with inadequately controlled blood pressure willing to participate, as well as more specific knowledge on the needed number of practices included, making the final sample size calculation uncertain at this point.

Randomisation Participating GPs will be randomly divided into two groups A and B, using the randomisation tool built into REDCap.

Participants will be given unique Trial Participant Numbers (TPNs). TPNs will be generated by PREDICT (the software behind Your Heart Forecast) when patients are included and will be given consecutively starting from 0001. The number will be given a prefix A or B depending on which group (intervention or control) the participant's general practice belongs to. Subgroup Q will be 5-15 participants chosen deliberately from the pilot group, to ensure it represents the intervention group for use in the qualitative interviews.

Practical procedure General practices will be actively involved in the RCT as follows. After identifying the list of patients from the statistics module, the practice will review the patients with regards to the inclusion/exclusion criteria. After reviewing, an invitational letter will be sent out to the first 25 of the remaining patients on the list. The invited patients can then opt out or show up at the appointment and receive the oral and written trial participant information. Patients will not need to go to the practice more times than usual, but the practice will need to use extra time to give trial information. The practice will be compensated for this extra time used.

The day after the inclusion, the participant will receive an email with a link to a questionnaire, which must be completed before the subsequent appointment with the GP. The first page of the questionnaire will be the informed consent form.

With the large number of patients with known hypertension and the compressed method of inclusion, it is expected that GPs will have enough use of the program Your Heart Forecast, to maintain the skills and knowledge to use the program, which they will be taught by the research group before inclusion.

The RCT will consist of a 12-month intervention period, except for participants in subgroup Q who will be interviewed 6 months after enrolment (t6) and subsequently excluded.

The intervention group will receive an educational e-mail, which also includes a reminder of the project and YHF, every 2 weeks. The e-mails' health educational content will reflect available information from the Danish Heart Association's web page (www.hjerteforeningen.dk).

Data:

The questionnaire (q1) will include questions to evaluate socioeconomic and sociodemographic variables, baseline health literacy, risk perception and self-efficacy (PAM-13), smoking status, comorbidity and medication.

The second patient questionnaire (q2) is very short and will focus on whether the patient was surprised about the risk score, if any changes in the medication were made and how the general experience of the YHF was.

Data regarding number and content of contacts to the GP will be obtained from the patient´s medical records and the affiliated accounting system including prescription databases for estimating compliance. All telephone-, email-, clinic- and home consultations are registered. Contacts from three years prior to the intervention and up until two years after, will be obtained.

Patients in the intervention group will receive their personal profile in the YHF to make it possible for them to access and use the program at home in between the blood pressure consultations at their GP. All data entered in YHF will be stored in accordance with Danish law by the software provider, with whom a data management agreement has been made.

Base-line measurements will be used to identify subgroups of participants. Qualitative data will be obtained via semi-structured interviews, transcribed and analysed with systematic text condensation. The qualitative interviews will seek to shed light on possible explanations for the hypothesized effects on self-management, lifestyle choices, blood pressure and contacts to the GP.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must understand and read Danish and must be cognitively well functioning.
2. The patient must have Internet access, host an email address and read their emails on regular basis (at least once a week).
3. Patients must give informed consent prior to inclusion.
4. All included patients must be diagnosed with hypertension and go to regular blood pressure control consultations at their GP (at least once a year).
5. Both patients with known hypertension and those newly discovered are accepted into the trial.
6. Age from 35 to 75 years (both included).
7. Both genders are included.
8. Comorbidity is allowed with a few exceptions (see exclusion criteria).

Exclusion Criteria:

1. If the patient during the trial, no longer fulfils inclusion criteria 1 and/or 2, they are excluded from the trial.
2. If the patient during the trial develops prolonged illness so severe that treatment of hypertension is no longer a priority, he/she will be excluded.
3. Patients with blood pressure above 170/100 are excluded, as these patients should receive intensive blood pressure treatment regardless of their predicted CVD risk or heart age.
4. Pregnancy.
5. Very high cholesterol (TCL or TCL/HDL 8 or over).
6. Genetic lipid disorders.
7. If the patient is diabetic AND has a complicating kidney disease.
8. Known problems with arteries to the legs defined as:

   1. Clinical symptoms of claudication
   2. Diminished foot pulses
   3. Carotid bruits
   4. Radiological evidence
   5. Prior surgery /percutaneous interventions
9. Prior stroke or mini-stroke (TIA).
10. Angina, prior AMI or heart related operation.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Health literacy | Questionnaire sent out at inclusion, after 6 months and after 1 year
  Self-reported change in health literacy through questionnaires.

SECONDARY OUTCOMES:
Blood pressure | Calculated after the 1 year trial period
  Difference in blood pressure from baseline to 1 year follow up consultation. Data will be put in the PREDICT project-database by the general practitioners.
Adherence | Questionnaire sent out at inclusion, after 6 months and after 1 year
  Change in adherence measured from prescription outtakes registered in the national prescription database and self-reported through questionnaire.
Empowerment | Questionnaire sent out at inclusion, after 6 months and after 1 year
  Empowerment measured with Patient Activation Measure 13 (PAM-13, Danish validated version) incorporated in the questionnaire (q1).
Number of contacts | Counted after end of 1 year trial period.
  Number and type of contacts from patient to doctor is counted and categorized. Data obtained from patient medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper B Nielsen, Professor, PhD, Study Chair — Research Unit of General Practice, University of Southern Denmark; Anders E Jensen, M.D., Principal Investigator — Research Unit of General Practice, University of Southern Denmark
Locations (1):
- Research Unit of General Practice, Department of Public Health, University of Southern Denmark, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Data from the project is only intended to be shared by publishing anonymised results.

REFERENCES:
- [Background] Reuther LO, Paulsen MS, Andersen M, Schultz-Larsen P, Christensen HR, Munck A, Larsen PV, Damsgaard J, Poulsen L, Hansen DG, Christensen B, Sondergaard J. Is a targeted intensive intervention effective for improvements in hypertension control? A randomized controlled trial. Fam Pract. 2012 Dec;29(6):626-32. doi: 10.1093/fampra/cms031. Epub 2012 May 7. PMID 22565110
- [Background] Soureti A, Hurling R, Murray P, van Mechelen W, Cobain M. Evaluation of a cardiovascular disease risk assessment tool for the promotion of healthier lifestyles. Eur J Cardiovasc Prev Rehabil. 2010 Oct;17(5):519-23. doi: 10.1097/HJR.0b013e328337ccd3. PMID 20195154
- [Background] Pedersen KM, Andersen JS, Sondergaard J. General practice and primary health care in Denmark. J Am Board Fam Med. 2012 Mar;25 Suppl 1:S34-8. doi: 10.3122/jabfm.2012.02.110216. PMID 22403249
- [Background] Brust-Renck PG, Royer CE, Reyna VF. Communicating Numerical Risk: Human Factors That Aid Understanding in Health Care. Rev Hum Factors Ergon. 2013 Oct;8(1):235-276. doi: 10.1177/1557234X13492980. PMID 24999307
- [Background] Berkman ND, Sheridan SL, Donahue KE, Halpern DJ, Crotty K. Low health literacy and health outcomes: an updated systematic review. Ann Intern Med. 2011 Jul 19;155(2):97-107. doi: 10.7326/0003-4819-155-2-201107190-00005. PMID 21768583
- [Background] Wells S, Kerr A, Eadie S, Wiltshire C, Jackson R. 'Your Heart Forecast': a new approach for describing and communicating cardiovascular risk? Heart. 2010 May;96(9):708-13. doi: 10.1136/hrt.2009.191320. No abstract available. PMID 20424153
- [Background] De Geest S, Sabate E. Adherence to long-term therapies: evidence for action. Eur J Cardiovasc Nurs. 2003 Dec;2(4):323. doi: 10.1016/S1474-5151(03)00091-4. No abstract available. PMID 14667488
- [Background] Maindal HT, Sokolowski I, Vedsted P. Translation, adaptation and validation of the American short form Patient Activation Measure (PAM13) in a Danish version. BMC Public Health. 2009 Jun 29;9:209. doi: 10.1186/1471-2458-9-209. PMID 19563630
- [Background] Sorensen K, Pelikan JM, Rothlin F, Ganahl K, Slonska Z, Doyle G, Fullam J, Kondilis B, Agrafiotis D, Uiters E, Falcon M, Mensing M, Tchamov K, van den Broucke S, Brand H; HLS-EU Consortium. Health literacy in Europe: comparative results of the European health literacy survey (HLS-EU). Eur J Public Health. 2015 Dec;25(6):1053-8. doi: 10.1093/eurpub/ckv043. Epub 2015 Apr 5. PMID 25843827
- [Background] Perestelo-Perez L, Rivero-Santana A, Boronat M, Sanchez-Afonso JA, Perez-Ramos J, Montori VM, Serrano-Aguilar P. Effect of the statin choice encounter decision aid in Spanish patients with type 2 diabetes: A randomized trial. Patient Educ Couns. 2016 Feb;99(2):295-9. doi: 10.1016/j.pec.2015.08.032. Epub 2015 Sep 1. PMID 26343571
- [Background] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Background] Madsbad S, Larsen ML, Adeler HF, Kryhlmand M, Westergaard M. [Implementation of clinical guidelines in general practice. The effect of journal audit and continuing education for the treatment of cardiovascular risk factors in patients with and without type 2 diabetes]. Ugeskr Laeger. 2006 Apr 24;168(17):1640-5. Danish. PMID 16674875
- [Derived] Stjernholm K, Andersen HS, Jensen AE, Nielsen JB. Danish evaluation of Your Heart Forecast: a cluster randomised controlled trial aimed at improving modifiable risk factors of CVD. Open Heart. 2026 Jan 28;13(1):e003812. doi: 10.1136/openhrt-2025-003812. PMID 41605571
- [Derived] Jensen AE, Sondergaard J, Kjaer NK, Jackson R, Nielsen JB. Danish Evaluation of Your Heart Forecast (DANY): study protocol for a cluster randomised controlled trial on an interactive risk-communication tool aimed at improving adherence of patients with high blood pressure. Trials. 2020 Jan 3;21(1):11. doi: 10.1186/s13063-019-3886-2. PMID 31900231